CLINICAL TRIAL: NCT01961271
Title: Multicentre Study To Evaluate Efficacy And Safety Of Buprenorphine Transdermal Patch (Norspan) In Chronic Non-Malignant Pain Of Moderate To Severe Intensity Due To Osteoarthritis, Rheumatoid Arthritis, Lower Back Pain And Joint / Muscle Pain, When Opioid Is Needed For Analgesia
Brief Title: Evaluation Of Efficacy And Safety Of Norspan In Moderate To Severe Pain Due To Osteoarthritis, Rheumatoid Arthritis, Joint/Muscle Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Pte Ltd. (Industry)
Collaborators: Mundipharma Korea Ltd (Industry); Mundipharma (Hong Kong) Ltd (Unknown); Mundipharma Distribution GmBH (Philippine Branch) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP12-AP-401
Record Dates: First submitted 2013-10-07; First posted 2013-10-11 (Estimated); Results first posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Lower Back Pain; Joint Pain; Muscle Pain
Keywords: Norspan; buprenorphine; transdermal; patch; chronic pain; non-malignant; osteoarthritis; rheumatoid arthritis; lower back pain; joint pain; muscle pain; opioid; analgesic; painkiller; Mundipharma
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Low Back Pain; Arthralgia; Myalgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Buprenorphine transdermal patch (Experimental): Subjects will be on either 5mg, 10mg, 15mg, 20mg, 25mg, 30mg or 40mg doses for 17 weeks. Dose titration will occur every week for the first 6 weeks, and will be maintained for the next 11 weeks.
  Interventions: Drug: Buprenorphine transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Please see Arm Description.
  Other Names: Norspan transdermal patch; Sovenor transdermal patch

SUMMARY:
The purpose of this study is to assess the efficacy of the buprenorphine transdermal patch (Norspan® or Sovenor® transdermal patch) in patients with chronic non-malignant pain of moderate to severe intensity due to osteoarthritis, rheumatoid arthritis, lower back pain and joint/muscle pain, who are not adequately responding to non-opioid painkillers.

DETAILED DESCRIPTION:
Baseline assessment (Visit 1) includes medical history, physical examination, vital signs.

At Visit 2 [7 days ( ± 3 days) after Visit 1] and subsequent optional titration visits up to (Visit 1 + 42 days) , patients will be titrated up to an effective and tolerated dose of Norspan® or Sovenor® transdermal patch and continue rescue analgesic, if necessary.

Titration period is dependent on time to achieving optimal pain control as determined by the investigator. The up-titration regime is planned on a weekly basis. Earlier dose titration (i.e. minimum 3 days after the patch application) is permitted at the investigator's discretion if the pain is uncontrolled. Effective and tolerated dose is assessed by data recorded in the case report form and patient diary.

According to country label, all patients will begin treatment with Norspan® or Sovenor® transdermal patch 5mg and will then be up-titrated, if necessary, to a maximum of Norspan® or Sovenor® transdermal patch 40mg or according to country label to achieve stable pain control. Patients that require oral opioid at any time during the study should be discontinued from the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-80 years (both inclusive) at the time of recruitment.
2. Clinical diagnosis of osteoarthritis, rheumatoid arthritis, lower back pain or joint / muscle pain.
3. Having non-malignant pain of moderate or severe intensity requiring an opioid for adequate analgesia (according to local label of Norspan® or Sovenor®). This is to be determined using BS-11 scores, where the cut-off point is ≥4.
4. Patients with chronic uncontrolled pain and is assessed to require opioid treatment but have not been treated with opioids (including tramadol, morphine etc.) within 4 weeks or more before study entry.

Exclusion Criteria:

1. Pregnant and lactating females.
2. Patients with chronic condition(s), in addition to osteoarthritis, that require(s) frequent analgesic treatment (e.g. frequent headaches, frequent migraine, and gout).
3. Patients who are awaiting a scheduled operation or other surgical procedure during study period or 3 months or less post-operative.
4. Prior history of being on opioids in the preceding 1 month prior to the study for the management of chronic non-malignant pain.
5. Prior history of buprenorphine transdermal system use.
6. Patients with history of allergic reactions against paracetamol/ acetaminophen, NSAIDs and/or opioids.
7. Patients with allergies or other contraindications to transdermal systems or patch adhesives.
8. Patients with dermatological disorders who may have problems applying patch or rotating patch placement area.
9. Patients with cancer (except for basal cell carcinoma) or history of cancer who have been diagnosed within five years prior to the first study visit (except for treated basal cell carcinoma).
10. Patients with conditions such as brain tumour, brain injury or raised intracranial pressure.
11. Patients with history of psychiatric disorder, uncontrollable epilepsy, untreated depression or other psychiatric disorders of a type that would make participation in the study an unacceptable risk to the patient.
12. Patients with any conditions causing poor cognitive function as assessed by the participating physician.
13. Patients with history of alcohol and drug abuse or patients who have demonstrated behaviour that suggests a dependency or drug abuse.
14. Patients currently taking hypnotics or other central nervous system depressants that may pose a risk of additional central nervous system depression with study medication.
15. Patients who are currently being administered monoamine oxidase inhibitors (MAOIs) or have taken MAOIs within 2 weeks before screening.
16. Patients requiring dose titration of adjuvant analgesics i.e. antidepressants (e.g. amitriptyline, amoxapine, clomipramine, selective serotonin re-uptake inhibitors (SSRIs)) and anticonvulsants (e.g. gabapentin, pregabalin). Patients will be allowed to enter the study as long as they are on the stable doses of adjuvant analgesics at screening and do not have dose adjustments during the study.
17. Patients who have received steroid treatment (intra-articular, intramuscular, oral, intravenous, epidural or other corticosteroid injections) within 6 weeks prior to clinical study or planned steroid treatment during the clinical study period.
18. Patients who have to use heating facility (examples: heating lamp, electric blanket, sauna, warm compresses, heated saline baths, etc.).
19. Patients who cannot or do not wish to remove hair growing at body surface where the patch can be placed.
20. Patients who are currently on disability claims or in the process of applying for disability claims.
21. Patients at child-bearing age who are planning to conceive a child during the study period and are not practicing adequate contraception.
22. Patients with known severe hepatic impairment as determined by liver function test within the past one year.
23. Patients who are currently in or have participated in other clinical trials within the last 30 days prior to study recruitment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- Hong Kong (6):
  - Pok Oi Hospital, Yuen Long, New Territories
  - Queen Elizabeth Hospital, Gascoigne Road
  - Queen Mary Hospital (Dept of Anaesthesiology), Pokfulam Road
  - Queen Mary Hospital (Dept of Rheumatology), Pokfulam Road
  - Prince of Wales Hospital, Shatin
  - Tuen Mun Hospital, Tuenmen
- Philippines (4):
  - Makati Medical Center, Makati City
  - Philippine General Hospital, Manila
  - University of Santo Tomas Hospital, Manila
  - St. Luke's Medical Center, Quezon City
- South Korea (6):
  - Samsung Medical Center, Gangnam-Gu, Seoul
  - Seoul National University Hospital (Dept of Neurology), Jongno-gu, Seoul
  - Seoul National University Hospital (Dept of Orthopedics), Jongno-gu, Seoul
  - Seoul St. Mary's Hospital, Seocho-gu, Seoul
  - Severance Hospital, Seodaemun-gu, Seoul
  - Asan Medical Center, Songpa-Gu, Seoul

REFERENCES:
- [Derived] Yoon DH, Bin SI, Chan SK, Chung CK, In Y, Kim H, Lichauco JJ, Mok CC, Moon YW, Ng TK, Penserga EG, Shin DA, You D, Moon H. Effectiveness and tolerability of transdermal buprenorphine patches: a multicenter, prospective, open-label study in Asian patients with moderate to severe chronic musculoskeletal pain. BMC Musculoskelet Disord. 2017 Aug 4;18(1):337. doi: 10.1186/s12891-017-1664-4. PMID 28778219

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buprenorphine Transdermal Patch
Started | 114
Completed | 64
Not Completed | 50

BASELINE CHARACTERISTICS:
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 28
Region of Enrollment [Number; unit: participants]
  Hong Kong | 26
  Philippines | 26
  Korea, Republic of | 62

OUTCOME MEASURES:

1. Primary Outcome: Efficacy According to BS-11 Pain Score Reduction
Description: The primary efficacy outcome analysis is the pre- and post-intervention change in BS-11 pain score. The reduction in scores were calculated by subtracting the post-intervention score from the baseline score.
  BS-11 is known as "Box scale-11"; it is an 11-point scale measuring pain intensity. It ranges from 0 to 10, whereby 0 represents no pain and 10 represents the worst imaginable pain. Subjects selected a number based on the pain intensity they were feeling at that time.
Time Frame: Maximum 17 weeks starting from enrolment
Population: Subjects of the analysis population met the eligibility criteria. It consists of subjects who completed the study and who withdrew for any reason.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 114
units on a scale | 2.7 (2.4)

2. Secondary Outcome: Secondary Efficacy Outcome Determined by Change in Percentage of Subjects Who Met Criteria on EQ5D-3L Quality of Life Questionnaire From Pre- to Post-intervention
Description: Pre-intervention: Visit 1 Post-intervention: Visit 6
  There are 5 dimensions in the EQ5D-3L questionnaire answered by the subjects, classified into 5 categories here:
  Mobility -- change in % of subjects who have no problem in walking around Self-care -- change in % of subjects who have no problem in self-care Usual activities -- change in % of subjects who have no problem with performing their usual activities Pain/ discomfort -- change in % of subjects who do not experience pain or discomfort Anxiety/ depression -- change in % of subjects who do not feel anxious or depressed
Time Frame: approximately 17 weeks starting from enrolment
Measure: Number; unit: percentage of subjects
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 114
percentage of subjects
  Mobility | 25.8
  Self-care | 20.2
  Usual Activities | 19.4
  Pain/Discomfort | 14.3
  Anxiety/ Depression | 18

3. Secondary Outcome: Treatment-emergent Adverse Events (TEAE's) as Measured by Number of Subjects With at Least 1 TEAE
Description: Side effects of the transdermal patch treatment will be analysed.
Time Frame: From time of enrolment up to 7 days after completion / discontinuation visit (up to 140 days)
Measure: Number; unit: participants
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 114
participants | 89

4. Secondary Outcome: Secondary Efficacy Outcome as Measured by Number of Subjects Requiring at Least 1 Breakthrough (Rescue) Pain Medication
Description: Daily use of breakthrough pain medication from visits 1-6, assessed from patient diaries.
Time Frame: Approximately 17 weeks starting from enrolment
Measure: Number; unit: participants
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 114
participants | 26

5. Secondary Outcome: Secondary Efficacy Outcome on Physicians' and Patients' Treatment Satisfaction Assessed Using Physician's Global Impression of Change Scale and Patient's Global Impression of Change Scale Respectively
Description: The overall assessment of the change in pain intensity from baseline is measured at Visit 6.
  Physician's Global Impression of Change scale: Investigator's opinion on a scale of 1 to 7 where 1 is "very much improved" and 7 is "very much worse" Patient's Global Impression of Change scale: Subject's opinion on a scale of 1 to 7 where 1 is "very much improved" and 7 is "very much worse"
Time Frame: At visit 6 (anywhere between Day 91 to 119 after enrolment depending on how long titration took)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 114
units on a scale
  Physician Impression | 2.62 (0.84)
  Patient Impression | 2.66 (0.81)

6. Secondary Outcome: Secondary Efficacy Outcome -- Incidence of Early Treatment Discontinuation Due to Lack of Efficacy.
Time Frame: From time of enrolment to Visit 6 (ie. up to119 days from enrolment)
Measure: Number; unit: participants
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 114
participants | 3

ADVERSE EVENTS:
Time Frame: The timeframe is up to 140 days. All adverse events will be recorded from the time the ICF is signed until 7 days after the completion/ discontinuation visit.
Arm/Group | Buprenorphine Transdermal Patch
Serious Adverse Events (participants affected / at risk) | 1/114
Other Adverse Events (participants affected / at risk) | 89/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine Transdermal Patch (N=114)
Hypertensive Crisis (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buprenorphine Transdermal Patch (N=114)
Atrial Tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Abdominal Discomfort (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 36
Diarrhea (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gingival Ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 45
Periodontitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 19
Application Site Erythema (General disorders) | 1
Application Site Irritation (General disorders) | 1
Application Site Pruritus (General disorders) | 5
Application Site Rash (General disorders) | 2
Application Site Swelling (General disorders) | 1
Application Site Warmth (General disorders) | 1
Asthenia (General disorders) | 2
Chest Discomfort (General disorders) | 1
Chest Pain (General disorders) | 1
Fatigue (General disorders) | 3
Feeling Cold (General disorders) | 1
Influenza-like Illness (General disorders) | 1
Edema (General disorders) | 1
Pyrexia (General disorders) | 1
Allergy to Arthropod Sting (Immune system disorders) | 1
Acute Tonsillitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Paronychia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Vaginal Infection (Infections and infestations) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Muscle Injury (Injury, poisoning and procedural complications) | 1
Muscle Strain (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 31
Headache (Nervous system disorders) | 10
Hypoesthesia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 22
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary Hesitation (Renal and urinary disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Cold Sweat (Skin and subcutaneous tissue disorders) | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertensive Crisis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data emerging from the study cannot be released without the permission of the sponsor.